CLINICAL TRIAL: NCT03096262
Title: Feasibility of a Kinect-Based Citizen Science Telerehabilitation Platform
Brief Title: Transforming Robot-mediated Telerehabilitation: Citizen Science for Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Science Foundation (Unknown); Foundation for Physical Medicine and Rehabilitation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: IRB00225650
Record Dates: First submitted 2017-03-24; First posted 2017-03-30 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Hemiparesis; Stroke
Keywords: cognitive skills; technical; internet platform; Stroke; Hemiparesis
MeSH Terms: conditions — Paresis; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stroke Patients (Experimental)
  Interventions: Device: Citizen Science intervention using kinect

INTERVENTIONS:
Device: Citizen Science intervention using kinect — Users are asked to tag objects on a screen

SUMMARY:
The purpose of this study is to advance upper limb robot-mediated tele-rehabilitation for patients recovering from stroke by empowering them through active science participation. By varying the tasks' features and affordances of a platform that combines a low-cost haptic device on one hand, and an online citizen science platform on the other, investigators will evaluate different strategies for social telerehabilitation. the two fundamental modes of social interaction - competition and cooperation - in addition to a control condition. Specifically, citizen science activities will be performed by competing, cooperating, or isolated users, and their rehabilitation effectiveness examined. Such effectiveness will be measured by (i) participants' rehabilitation performance (inferred from sensorimotor data acquired through the platform and directly quantified by a supervising therapist); (ii) participants' motivations to contribute (measured through surveys administered online); and (iii) participants' emotional well-being and sense of self-esteem (measured through online surveys).

ELIGIBILITY:
Inclusion Criteria:

For treatment group:

* post-stroke hemiparesis >3 months
* ability to stand or sit independently
* sufficient cognitive skills to perform the exercises as demonstrated
* full passive range of motion in the affected arm but limited active movement as determined by a upper extremity Fugl-Meyer score of <50/66
* technical savvy and interest to use an internet platform

For control group:

(ii) no history of learning disabilities (iii) technical savvy and interest to use an internet platform

Exclusion Criteria:

For treatment group:

* visual deficit such as deficit in visual acuity, eye movements, visual field cut, or neglect
* medical comorbidity such as other neurological conditions (e.g. Parkinson's disease, brain tumor, epilepsy), or previous injury to the upper limb
* pain in the upper limbs that prevents full passive range of motion to perform the exercises.

For control group:

* visual deficit such as deficit in visual acuity, eye movements, visual field cut, or neglect
* any previous injury or medical condition that prevents full passive range of motion to perform the exercises.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Feasibility of the kinect motion capture platform to capture movement assessed by range of motion | 1 day
  Range-of-motion measurements of the affected and unaffected arm using the kinect motion capture platform.
Feasibility of the kinect motion capture platform to capture workload assessed by NASA Task Load Index | 1 day
  Assesses work load on five 7-point scales. A series of measures that capture workload. Each scale employs a visual analog scale that measures each of the domains. The domains are Mental Domain, Physical Demand, Temporal Demand, Performance, Effort and Frustration Level. Each scale domain and the Composite has a range from 0 to 100 with 100 being the highest indicator of workload.
Feasibility of the kinect motion capture platform usability assessed by the System usability scale | 1 day
  Using a 10 item scale to assess the usability of the technology platform with stroke patients. The measure is scored on a 0-100 scale, a higher score means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Preeti Raghavan, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Matthew Bird, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No